CLINICAL TRIAL: NCT03120442
Title: Postoperative Delirium After Total Knee Arthroplasty Under Regional Anesthesia: a Comparison Between Intraoperative Sedation With Fentanyl, Fentanyl-dexmedetomidine and Fentanyl-propofol
Brief Title: Postoperative Delirium After Total Knee Arthroplasty Under Regional Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, patcharee sriswasdi, MD, MPH, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 051/2560(EC2)
Record Dates: First submitted 2017-04-15; First posted 2017-04-19 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Delirium
Keywords: postoperative delirium; total knee arthroplasty; propofol; dexmedetomidine; fentanyl; inflammatory response; interleukins; CAM-ICU
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol; Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol-fentanyl (Experimental): Fentanyl 0.5 mcg/kg Propofol Target-controlled infusion to achieve MOAA/S 3-4 as end point of sedation Bispectral index (BIS) monitoring
  Interventions: Drug: Propofol; Drug: Fentanyl
- Dexmedetomidine (Experimental): Fentanyl 0.5 mcg/kg Dexmedetomidine in incremental titrated dose for moderate sedation to achieve MOAA/S 3-4 as end-point of titration Bispectral index (BIS) monitoring
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl
- Fentanyl (Experimental): Fentanyl 0.5 mcg/kg Supplemental dosage of fentanyl for intraoperative anxiolysis
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Propofol — target-controlled infusion starting for Cet 0.1 mcg/ml to achieve MOAA/S 3-4
  Arms: Propofol-fentanyl
Drug: Dexmedetomidine — Incremental titration of dexmedetomidine starting from 0.1 mcg/kg/hr to achieve MOAA/S 3-4
  Arms: Dexmedetomidine
Drug: Fentanyl — 0.25 mcg fo Fentanyl for anxiolysis

SUMMARY:
Postoperative delirium after total knee replacement surgery has been related to significant morbidity and mortality among high risk patients. Anesthetic care might play a role in the development of postoperative delirium.

The purpose of this study is to compare the incidence of postoperative delirium between different intraoperative sedation regimen. Delirium assessment using standardized screening tools will be done every 8 hours after surgery.

DETAILED DESCRIPTION:
* In this randomized controlled trial, the investigator will compare the incidence of postoperative delirium after total knee arthroplasty between 3 intraoperative sedation regimens including (1) propofol-fentanyl (2) dexmedetomidine -fentanyl (3) fentanyl alone
* Anesthesia techniques include spinal anesthesia and adductor canal block for postoperative analgesia. Sedation will be provide per group assignment.
* After performance of regional anesthesia, sedation protocols will be used as followed: (1) target-controlled infusion of Propofol to achieve MOAA/S of 3-4 (2) incremental titration of Dexmedetomidine to achieve MOAA/S of 3-4 (3) supplemental fentanyl for anxiolysis.
* Delirium will be screened by trained physicians, registered nurses every 8 hours postoperatively with validated Thai-version CAM-ICU (Confusion Assessment Method-Intensive Care Unit) until patient discharge.
* Serum Interleukins (IL-1, IL-6) Tumor necrosis factor-Alpha and S100B protein from preoperative period will be compared with serum from postoperative period between delirium and non-delirium group. The level of serum biomarkers will be acquired in a 6-hour interval for 5 measurement points during the first postoperative day in the first 12 participants. The subsequent participants will have 1 measurement of serum biomarker during the first postoperative day.
* Genetic profile for ApolipoproteinE genotype will be acquired and compared between delirium and non-delirium group.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 year or older
* Scheduled for elective primary total knee arthroplasty

Exclusion Criteria:

* Contraindication for spinal anesthesia
* Contraindication for adductor canal block
* Allergy to fentanyl or propofol or dexmedetomidine or bupivacaine
* Cognitive impairment
* NSQIP database risk calculator > 10% overall complication
* Unable to communicate in Thai language
* Significant visual and hearing impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium

SECONDARY OUTCOMES:
The effect of age on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between age 65-75, 75-85, and >85 years of age
Apolipoprotein genotype | 1 days
  ApoE epsilon subtype analysis
The effect of Apolipoprotein genotype on the incidence of postoperative delirium | Up to 7 days
  ApoE epsilon subtype analysis
Inflammatory biomarker | 2 days
  Preoperative and postoperative comparison of inflammatory biomarker (IL-1, IL-6 TNF, S100b protein)
The effect of delirium on inflammatory biomarker levels | Up to 7 days
  Preoperative and postoperative comparison of inflammatory biomarker (IL-1, IL-6 TNF, S100b protein) comparison between delirium and non-delirium group
The effect of gender on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between male and female
The effect of ASA-physical status on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between ASA-PS I-II and III-IV
The effect of alcohol consumption on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between amount of alcohol consumption (standard drink/day)
The effect of cognitive inpairment on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between patients with and without cognitive impairment. TMSE score will be use to determine cognitive status
The effect of coronary artery disease on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between patients with and without coronary artery disease. Preoperative diagnosis of coronary artery disease will be used.
The effect of cerebrovascular disease on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between patients with and without cerebrovascular disease. Preoperative diagnosis of cerebrovascular disease will be used.
The effect of chronic kidney disease on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between patients with and without chronic kidney disease. Preoperative diagnosis of cerebrovascular disease will be used.
The effect of liver disease on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between patients with and without liver disease. Preoperative diagnosis of liver disease will be used.
The effect of hypertension on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between patients with and without hypertension. Preoperative diagnosis of hypertension will be used.
The effect of diabetes mellitus on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between patients with and without diabetes mellitus. Preoperative diagnosis of diabetes will be used.
The effect of postoperative pain on the incidence of postoperative delirium | Up to 7 days
  Positive CAM-ICU result and confirmed DSM-V criteria for delirium between patients with mild (pain score 0-3), moderate (4-7) and severe (7-10). Numeric rating scale will be used.
The effect of intraoperative BIS value on the incidence of postoperative delirium | 7 days
  Intraoperative BIS value comparison between delirium and non-delirium group. Positive CAM-ICU result and confirmed DSM-V criteria will be used to diagnose delirium
The effect of intraoperative blood transfusion and blood loss on the incidence of postoperative delirium | 7 days
  Intraoperative blood transfusion and blood loss will be compared between delirium and non-delirium group. Positive CAM-ICU result and confirmed DSM-V criteria will be used to diagnose delirium
The effect of delirium on hospital length of stay | 7 days
  The hospital length of stay will be compared between delirium and non-delirium group. Positive CAM-ICU result and confirmed DSM-V criteria will be used to diagnose delirium
The effect of delirium on postoperative rehabilitation | 7 days
  The time to assisted walking in the postoperative period will be compared between delirium and non-delirium group. Positive CAM-ICU result and confirmed DSM-V criteria will be used to diagnose delirium
The effect of delirium on postoperative complications. | 7 days
  The incidence of 1) DVT 2) myocardial ischemia/infarction 3) urinary tract infection 4) stroke 5) wound infection will be compared between delirium and non-delirium group. Positive CAM-ICU result and confirmed DSM-V criteria will be used to diagnose delirium

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gleason LJ, Schmitt EM, Kosar CM, Tabloski P, Saczynski JS, Robinson T, Cooper Z, Rogers SO Jr, Jones RN, Marcantonio ER, Inouye SK. Effect of Delirium and Other Major Complications on Outcomes After Elective Surgery in Older Adults. JAMA Surg. 2015 Dec;150(12):1134-40. doi: 10.1001/jamasurg.2015.2606. PMID 26352694
- [Background] da Silva RR, Santos AA, de Sampaio Carvalho Junior J, Matos MA. Quality of life after total knee arthroplasty: systematic review. Rev Bras Ortop. 2014 Sep 19;49(5):520-7. doi: 10.1016/j.rboe.2014.09.007. eCollection 2014 Sep-Oct. PMID 26229855
- [Background] Rade MC, Yadeau JT, Ford C, Reid MC. Postoperative delirium in elderly patients after elective hip or knee arthroplasty performed under regional anesthesia. HSS J. 2011 Jul;7(2):151-6. doi: 10.1007/s11420-011-9195-2. Epub 2011 Feb 11. PMID 22754416
- [Background] Kinjo S, Lim E, Sands LP, Bozic KJ, Leung JM. Does using a femoral nerve block for total knee replacement decrease postoperative delirium? BMC Anesthesiol. 2012 Mar 10;12:4. doi: 10.1186/1471-2253-12-4. PMID 22405052
- [Background] Yen TE, Allen JC, Rivelli SK, Patterson SC, Metcalf MR, Flink BJ, Mirrakhimov AE, Lagoo SA, Vail TP, Young CC, Moon RE, Trzepacz PT, Kwatra MM. Association between Serum IGF-I levels and Postoperative Delirium in Elderly Subjects Undergoing Elective Knee Arthroplasty. Sci Rep. 2016 Feb 5;6:20736. doi: 10.1038/srep20736. PMID 26846868
- [Background] Liang CK, Chu CL, Chou MY, Lin YT, Lu T, Hsu CJ, Chen LK. Interrelationship of postoperative delirium and cognitive impairment and their impact on the functional status in older patients undergoing orthopaedic surgery: a prospective cohort study. PLoS One. 2014 Nov 17;9(11):e110339. doi: 10.1371/journal.pone.0110339. eCollection 2014. PMID 25402484
- [Background] Liang CK, Chu CL, Chou MY, Lin YT, Lu T, Hsu CJ, Lam HC, Chen LK. Developing a Prediction Model for Post-Operative Delirium and Long-Term Outcomes Among Older Patients Receiving Elective Orthopedic Surgery: A Prospective Cohort Study in Taiwan. Rejuvenation Res. 2015 Aug;18(4):347-55. doi: 10.1089/rej.2014.1645. PMID 25768947
- [Background] Nandi S, Harvey WF, Saillant J, Kazakin A, Talmo C, Bono J. Pharmacologic risk factors for post-operative delirium in total joint arthroplasty patients: a case-control study. J Arthroplasty. 2014 Feb;29(2):268-71. doi: 10.1016/j.arth.2013.06.004. Epub 2013 Jul 5. PMID 23831083
- [Background] Scott JE, Mathias JL, Kneebone AC. Incidence of delirium following total joint replacement in older adults: a meta-analysis. Gen Hosp Psychiatry. 2015 May-Jun;37(3):223-9. doi: 10.1016/j.genhosppsych.2015.02.004. Epub 2015 Feb 23. PMID 25774049
- [Background] Vasunilashorn SM, Ngo L, Inouye SK, Libermann TA, Jones RN, Alsop DC, Guess J, Jastrzebski S, McElhaney JE, Kuchel GA, Marcantonio ER. Cytokines and Postoperative Delirium in Older Patients Undergoing Major Elective Surgery. J Gerontol A Biol Sci Med Sci. 2015 Oct;70(10):1289-95. doi: 10.1093/gerona/glv083. Epub 2015 Jul 27. PMID 26215633
- [Background] Fournier A, Krause R, Winterer G, Schneider R. Biomarkers of postoperative delirium and cognitive dysfunction. Front Aging Neurosci. 2015 Jun 9;7:112. doi: 10.3389/fnagi.2015.00112. eCollection 2015. PMID 26106326
- [Background] Peng L, Xu L, Ouyang W. Role of peripheral inflammatory markers in postoperative cognitive dysfunction (POCD): a meta-analysis. PLoS One. 2013 Nov 13;8(11):e79624. doi: 10.1371/journal.pone.0079624. eCollection 2013. PMID 24236147
- [Background] Tomaszewski D. Biomarkers of Brain Damage and Postoperative Cognitive Disorders in Orthopedic Patients: An Update. Biomed Res Int. 2015;2015:402959. doi: 10.1155/2015/402959. Epub 2015 Aug 31. PMID 26417595
- [Background] Hirsch J, Vacas S, Terrando N, Yuan M, Sands LP, Kramer J, Bozic K, Maze MM, Leung JM. Perioperative cerebrospinal fluid and plasma inflammatory markers after orthopedic surgery. J Neuroinflammation. 2016 Aug 30;13(1):211. doi: 10.1186/s12974-016-0681-9. PMID 27577265
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] van Munster BC, Bisschop PH, Zwinderman AH, Korevaar JC, Endert E, Wiersinga WJ, van Oosten HE, Goslings JC, de Rooij SE. Cortisol, interleukins and S100B in delirium in the elderly. Brain Cogn. 2010 Oct;74(1):18-23. doi: 10.1016/j.bandc.2010.05.010. Epub 2010 Jun 26. PMID 20580479
- [Background] Krenk L, Rasmussen LS, Hansen TB, Bogo S, Soballe K, Kehlet H. Delirium after fast-track hip and knee arthroplasty. Br J Anaesth. 2012 Apr;108(4):607-11. doi: 10.1093/bja/aer493. Epub 2012 Jan 24. PMID 22277666
- [Background] Krenk L, Kehlet H, Baek Hansen T, Solgaard S, Soballe K, Rasmussen LS. Cognitive dysfunction after fast-track hip and knee replacement. Anesth Analg. 2014 May;118(5):1034-40. doi: 10.1213/ANE.0000000000000194. PMID 24781572
- [Background] Orena EF, King AB, Hughes CG. The role of anesthesia in the prevention of postoperative delirium: a systematic review. Minerva Anestesiol. 2016 Jun;82(6):669-83. Epub 2016 Jan 28. PMID 26822815
- [Background] Djaiani G, Silverton N, Fedorko L, Carroll J, Styra R, Rao V, Katznelson R. Dexmedetomidine versus Propofol Sedation Reduces Delirium after Cardiac Surgery: A Randomized Controlled Trial. Anesthesiology. 2016 Feb;124(2):362-8. doi: 10.1097/ALN.0000000000000951. PMID 26575144
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Liu Y, Ma L, Gao M, Guo W, Ma Y. Dexmedetomidine reduces postoperative delirium after joint replacement in elderly patients with mild cognitive impairment. Aging Clin Exp Res. 2016 Aug;28(4):729-36. doi: 10.1007/s40520-015-0492-3. Epub 2015 Nov 11. PMID 26559412
- [Background] Sieber FE, Zakriya KJ, Gottschalk A, Blute MR, Lee HB, Rosenberg PB, Mears SC. Sedation depth during spinal anesthesia and the development of postoperative delirium in elderly patients undergoing hip fracture repair. Mayo Clin Proc. 2010 Jan;85(1):18-26. doi: 10.4065/mcp.2009.0469. PMID 20042557
- [Background] Chan MT, Cheng BC, Lee TM, Gin T; CODA Trial Group. BIS-guided anesthesia decreases postoperative delirium and cognitive decline. J Neurosurg Anesthesiol. 2013 Jan;25(1):33-42. doi: 10.1097/ANA.0b013e3182712fba. PMID 23027226
- [Background] Radtke FM, Franck M, Lendner J, Kruger S, Wernecke KD, Spies CD. Monitoring depth of anaesthesia in a randomized trial decreases the rate of postoperative delirium but not postoperative cognitive dysfunction. Br J Anaesth. 2013 Jun;110 Suppl 1:i98-105. doi: 10.1093/bja/aet055. Epub 2013 Mar 28. PMID 23539235
- [Background] Ely EW, Girard TD, Shintani AK, Jackson JC, Gordon SM, Thomason JW, Pun BT, Canonico AE, Light RW, Pandharipande P, Laskowitz DT. Apolipoprotein E4 polymorphism as a genetic predisposition to delirium in critically ill patients. Crit Care Med. 2007 Jan;35(1):112-7. doi: 10.1097/01.CCM.0000251925.18961.CA. PMID 17133176
- [Background] Leung JM, Sands LP, Wang Y, Poon A, Kwok PY, Kane JP, Pullinger CR. Apolipoprotein E e4 allele increases the risk of early postoperative delirium in older patients undergoing noncardiac surgery. Anesthesiology. 2007 Sep;107(3):406-11. doi: 10.1097/01.anes.0000278905.07899.df. PMID 17721242
- [Background] Cai Y, Hu H, Liu P, Feng G, Dong W, Yu B, Zhu Y, Song J, Zhao M. Association between the apolipoprotein E4 and postoperative cognitive dysfunction in elderly patients undergoing intravenous anesthesia and inhalation anesthesia. Anesthesiology. 2012 Jan;116(1):84-93. doi: 10.1097/ALN.0b013e31823da7a2. PMID 22108393
- [Background] Ward A, Crean S, Mercaldi CJ, Collins JM, Boyd D, Cook MN, Arrighi HM. Prevalence of apolipoprotein E4 genotype and homozygotes (APOE e4/4) among patients diagnosed with Alzheimer's disease: a systematic review and meta-analysis. Neuroepidemiology. 2012;38(1):1-17. doi: 10.1159/000334607. Epub 2011 Dec 17. PMID 22179327
- [Background] Gusmao-Flores D, Salluh JI, Chalhub RA, Quarantini LC. The confusion assessment method for the intensive care unit (CAM-ICU) and intensive care delirium screening checklist (ICDSC) for the diagnosis of delirium: a systematic review and meta-analysis of clinical studies. Crit Care. 2012 Jul 3;16(4):R115. doi: 10.1186/cc11407. PMID 22759376
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Pipanmekaporn T, Wongpakaran N, Mueankwan S, Dendumrongkul P, Chittawatanarat K, Khongpheng N, Duangsoy N. Validity and reliability of the Thai version of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Clin Interv Aging. 2014 May 29;9:879-85. doi: 10.2147/CIA.S62660. eCollection 2014. PMID 24904208